CLINICAL TRIAL: NCT04475172
Title: Evaluation Of Clinical Performance of Self-adhering Flowable Composite vs Conventional Flowable Composite in Cervical Carious Lesions: A Randomized Clinical Trial
Brief Title: Evaluation Of Clinical Performance of Self-adhering Flowable Composite vs Conventional Flowable Composite in Cervical Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatheya Mansour Atifa Elshnawy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECPSAFCsCFC
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fusio™ Flowable Self-Adhesive Flowable Composite (Experimental): 2-Cavity preparation steps:
  * patients will be given local anesthesia as required,the operative field will be isolated with rubber dam before starting.
  * Conventional design Class V cavity will be prepared on the buccal surface of tooth by No. #330 bur (0.8 mm in diameter and 1.6 mm in length) , tooth surfaces will be kept moist to protect them against dehydration.
  * 2% chlorhexidine gluconate disinfecting solution .
  * wash the dentin surface with water spray and air dry with maximum air pressure for 5 s.
  A) Intervention: Fusio™ Flowable (Self adhesive flowable composite):
  * Simply syringe into the preparation 1 mm increments, agitate with tip or brush for 20 s, and light-cure.No need for an etchant or an adhesive.
  Interventions: Combination Product: Self-Adhesive Flowable Composite
- Conventional flowable composite [Tetric Evo Flow (FF)]. (Active Comparator): Tetric Evo Flow (Conventional flowable composite):
  * After cleaning cavities, apply conditioning material (phosphoric acid etching 37% ) and apply bonding agent (ExciTE® F) according to the instructions for use of the product.
  * Apply Tetric EvoFlow in layers of 1mm. Polymerize each layer separately following the instructions for use of this product. . Hold the light emission window as closely as possible to the surface of the restorative material.
  All 20 Class V restorations will be prepared, restored, finished, and polished by one operator. Each of the 10 patients had one (FL) restoration and the other restoration will be filled with (FF).
  Interventions: Combination Product: Self-Adhesive Flowable Composite

INTERVENTIONS:
Combination Product: Self-Adhesive Flowable Composite — Fusio Self-Adhesive Flowable Composite combines the benefits of adhesive and restorative technology into one product . Immediately upon application Fusio conditions, bonds, and seals without the need for an etchant or an adhesive.
  It is based on the bonding technology that uses glycerophosphate dimethacrylate(GPDM)to etch enamel and dentin, and hydroxyethyl methacrylate (HEMA) to enhance wetting and penetration by resin into dentin.
  Other Names: Fusio™ Flowable Self-Adhesive Flowable Composite

SUMMARY:
This clinical trial will be conducted to compare the clinical performance of a new self-adhering flowable composite in restoring CLs compared to conventional flowable composite in geriatric patients over 12 months.

DETAILED DESCRIPTION:
Recently, self-adhesive flowable composites (SAFCs) have been introduced as a new class of restorative material in adhesive dentistry. Today, there are only two available products in the market for clinical use: Vertise Flow and Fusio Liquid Dentin. Self-adhering flowable composite was introduced to address the time-consuming procedure used with traditional materials Their resin matrix contains acidic functional adhesive monomers mediating bonding with dental hard tissues and, therefore, separate etching and additional bonding are not required. SAFCs have been mainly advertised for the restoration of small Class I, Class III and V cavities, for cavity lining, and for use as a pit and fissure sealant.

Self-adhering flowable composite combines the merits of both adhesive and restorative material technologies in one product, bringing novel horizons to restorative techniques, as it is a direct composite resin restorative material that has an adhesive resin together with a flowable composite resin. It is based on the bonding technology that uses glycerophosphate dimethacrylate(GPDM)to etch enamel and dentin, and hydroxyethyl methacrylate (HEMA) to enhance wetting and penetration by resin into dentin. This resin bonds chemically between the phosphate groups of a GPDM monomer and the hydroxyapatite of tooth structure and, also, micromechanically between the polymerized monomers of the self-adhering flowable composite resin and the collagen fibers and smear layer of dentin.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Class V carious lesions in anterior and premolars teeth.
* Age above 60 years.
* Males and females.

Exclusion Criteria:

* • patient less than 60 years with disabilities, systemic disease, severe medical conditions, rampant caries, and xerostomia.

  * In addition, teeth with potential prosthodontics restoration and nonvital or endodontically treated teeth.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Marginal integrity of Class V restorations | Clinical Evaluation of Marginal integrity after 6 months after starting treatment.
  clinical evaluation according to Modified USPHS Criteria (Bayne and Schmalz, 2005) unit of measurement :Alfa, Bravo,charlie and Delta

SECONDARY OUTCOMES:
Postoperative sensitivity | at baseline and 3 months after starting treatment .
  clinical evaluation according to Modified United States Public Health Service Criteria (Bayne and Schmalz, 2005)